CLINICAL TRIAL: NCT05803876
Title: Cerebral Perfusion Variation During Blood Pressure Changes Under General Anesthesia: Relationship Between Transcranial Doppler, Frontal EEG, and Cerebral Oximetry: a Prospective Observational Study
Brief Title: Cerebral Perfusion Variation During Blood Pressure Changes Under General Anesthesia
Acronym: DELTAPAMAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); M3DISIM (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230072; 2022-A02647-36 (Other: IDRCB)
Record Dates: First submitted 2023-03-16; First posted 2023-04-07 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: General Anesthesia
Keywords: Cerebrovascular Autoregulation; neurovascular coupling; Individualized vs Standard Blood Pressure Management Strategies; Multimodal monitoring; Brain Oxygen Saturation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General anesthesia: Patients undergoing surgery under general anesthesia with an intravenous anesthesia protocol with a concentration target (Orchestra® Base Primea - Fresenius Kabi France), a vasopressor support by norepinephrine and blood pressure optimisation.
  Interventions: Other: Diagnostic test - monitoring

INTERVENTIONS:
Other: Diagnostic test - monitoring — Continuous measurement of blood velocity in the middle cerebral artery by transcranial pulsed Doppler (TCD) Atys Medical TCD-X®. The probe attachment system on the patient's head looks like a pair of glasses; it is light and comfortable. The orientation of the robotic probe is automatically readjusted to ensure stable recording quality over time. (recorded on Data Warehouse Connect).
  For all patients Vm in (cm/s) will be collected during the adjustment of the mean arterial pressure level between 90% and 70% of the baseline value, without ever going below 60 mmHg for the patients at low risk and 80 mmHg for the patients at high cardiovascular risk.
  Other Names: Non-invasive measurement of cerebral blood velocity in the middle cerebral artery by transcranial pulsed Doppler (TCD) (Mean velocity, Vm, cm/s)

SUMMARY:
The risk associated with arterial hypotension during general anesthesia for surgery has been demonstrated , but the threshold at which consequences for perfusion of one or more organs appear varies according to the mechanism of hypotension, associated abnormalities (HR, cardiac output, and oxygen transport), and the patient's terrain.

Currently, a mean arterial pressure greater than 60 mm Hg and a reduction of less than 30-50% from the value measured before general anesthesia are commonly used treatment thresholds to ensure good perfusion of all organs.

Normally, cerebral blood flow is auto-regulated, which allows cerebral blood flow to adapt to oxygen requirements and to different levels of blood pressure, both high and low. However, this protective mechanism may fail for a degree of hypotension that depends on several factors such as the age or vascular status of the patient.

The aim of the study is to measure non-invasively, easily and reliably the variations of cerebral perfusion in patients with and without cardiovascular risk factors during controlled variations performed during routine care to set the blood pressure level within the recommended safety standards during general anesthesia.

What is the target level of blood pressure tolerable for a patient under general anesthesia? Is there a simple and non-invasive way to measure the level of cerebral blood flow autoregulation and especially its adequacy to the brain's oxygen needs?

DETAILED DESCRIPTION:
The risk associated with arterial hypotension during general anesthesia for surgery or interventional procedure has been demonstrated, but the threshold at which consequences for perfusion of one or more organs appear varies according to the mechanism of hypotension, associated abnormalities (Heart rate, cardiac output, and oxygen transport), and the patient's terrain.

Currently, a mean arterial pressure greater than 60 mm Hg and a reduction of less than 30-50% from the value measured before general anesthesia are commonly used treatment thresholds to ensure good perfusion of all organs.

These values are based on large cohort studies that associate these blood pressure thresholds with the occurrence of postoperative complications or during the resuscitation stay. They cannot be generalized to certain subpopulations that are underrepresented, such as women and elderly patients.

Normally, cerebral blood flow is self-regulated, which allows cerebral blood flow to adapt to oxygen requirements and to different levels of high and low blood pressure.

However, this protective mechanism may fail for a degree of hypotension that depends on several factors such as the age or vascular health of the patient. For example, in patients with preexisting hypertension, the autoregulatory capacity of the brain is likely impaired making organs more susceptible to ischemia at low blood pressure.

Thus, current American College of Cardiology and American Heart Association guidelines in the setting of noncardiac surgery recommend individualizing care for patients with associated cardiovascular comorbidities. Arterial stiffness is currently one of the best independent, early biomarkers predictive of cardiovascular complications and cardiovascular comorbidity. Assessment of arterial stiffness is currently performed by pulse wave velocity (PWV) measurement. Therefore, higher blood pressure goals tailored to the physiology of each patient may be preferable for these high-risk patients.

Because there is individual variability in cerebral autoregulation, a strategy based on a "one-size-fits-all" recommended blood pressure (BP) value is nonsense.

What is the tolerable target BP level for a patient under general anesthesia? Is there a simple and non-invasive way to measure the level of cerebral blood flow autoregulation and, more importantly, adequacy to the brain's oxygen requirements?

The aim of the study is to measure non-invasively, easily and reliably the variations of cerebral perfusion in patients with or without cardiovascular risk factors during controlled variations performed during routine care to adjust the blood pressure level within the recommended safety standards during general anesthesia. The setting of the optimal mean arterial pressure (MAP) level will be achieved within the ranges of values commonly used, taking into account the patient's cardiovascular comorbidities. In particular, the lower limit of MAP of 60 mmHg for patients without cardiovascular risk factors and 80 mmHg for patients with risk factors should never be exceeded, in accordance with current French and international recommendations. The main objective is to identify a significant linear relationship between the percentage change in mean velocity (Vm) and the percentage change in the 95% spectral frequency front (SEF95) during the MAP change.

Cerebral perfusion and cerebral O2 adequacy will be compared and assessed by continuous and simultaneous measurements of cerebral blood flow by transcranial Doppler (TCD) and cerebral O2 adequacy by near-infrared spectroscopy (NIRS) and a brain function parameter by intraoperative electroencephalogram (EEG) - frontal EEG.

The classification of patients in the cardiovascular risk group will be determined in addition to their history and treatment by an arterial stiffness parameter (pulse wave velocity) measured non-invasively before and during the protocol by MESI mTablet automatic digital sphygmomanometer (MESI ltd, Slovenia).

The objective for a given patient is to look for a possible threshold value of pressure that could impact the blood flow velocity (Doppler) and possibly the EEG and cerebral oximetry.

This clinical research work is performed on adult patients undergoing scheduled surgery at Lariboisière Hospital under general anaesthesia.

All measurements are obtained non-invasively. The monitoring routinely includes continuous electrocardiogram and blood pressure monitoring by non-invasive means (Clearsight®, EV1000®, Edwards Sciences) in anesthesia pulsed O2 saturation (SpO2), ventilatory parameters (FR, VC, FiO2), and anesthesia depth by frontal EEG.

Patients over 18 years of age are eligible to participate in this protocol. During the anaesthesia consultation, they will be given an information letter on the objectives and the course of the study. Their non-objection to participate in this study will be collected at the latest during the pre-anesthetic visit, the day before the operation, after a period of reflection. The protocol starts on the day of the operation.

For all patients, the surgical procedures will be performed under general anesthesia with an intravenous anesthesia protocol with a concentration target (Orchestra® Base Primea - Fresenius Kabi France) and a vasopressor support by norepinephrine diluted to 5 microg/mL. Blood pressure variations will be performed as follows:

In current practice of investigators :

* anesthetic induction is performed under vasopressors (norepinephrine diluted to 5 µg/mL) with the objective of maintaining a MAP ≥ 90% of the value measured during the anesthesia consultation.
* when blood pressure stability is obtained, the dose of norepinephrine is gradually decreased to a MAP target ≥ 70% of the baseline value without ever falling below 60 mmHg for patients without low cardiovascular risk factors and 80 mmHg for patients with cardiovascular risk factors.

At this stage the data to establish the autoregulatory threshold are not yet analyzed and are not available to adjust the mean arterial pressure level.

The change in cerebral blood flow will then be compared with the change in mean arterial pressure (dPAM) to obtain the slope of the change in mean velocity (dVm) of the blood in the middle cerebral artery obtained by transcranial Doppler (dVm/dPAM in percentage). In case of a positive correlation between these two parameters, cerebral autoregulation will be considered as impaired, and in case of no correlation it will be considered as preserved.

On the day of the intervention, a routine monitoring of the depth of anesthesia from the quantitative frontal EEG (Sedline Masimo®) ensures a continuous recording of the intraoperative EEG data. Placement of a frontal O3® Sensor rSO2 Masimo® or Foresight sensor rSO2 Edwards® electrode for continuous measurement of cerebral tissue O2 saturation (StO2). Continuous measurement of blood velocity in the middle cerebral artery by transcranial pulsed Doppler (TCD) Atys Medical TCD-X®. The probe attachment system on the patient's head is similar to a pair of glasses; it is light and comfortable. The orientation of the robotic probe is automatically readjusted to ensure stable recording quality over time.

Patients over 18 years old are eligible to participate in this protocol.

No additional examinations will be performed. The physician in charge of the study collecting the data is not involved in the patient's management at any time.

The monitoring data are currently available and are made available in the clinical research unit of department thanks to

* A data extraction system from the PHILIPS IntelliVue monitoring solutions. The Data Warehouse Connect software solution allows the collection of all these data with a fine sampling (2ms for the tracings, 1s for the numerical data), which considerably widens the capacities in terms of data analysis and exploitation.
* The retrieval system is temporally coupled to the patient's events, medications (doses) administered through an IntelliSpace Critical Care and Anesthesia (ICCAA) information system that is operational in all operating rooms. The clinical information system is linked to all medical devices and is fed by nurses to record events and the administration of medications and solutions. Thus, the data provided are coupled with the digital traces and measurements of the multiparametric monitor, transmitted in HL7 to the server of the hospital's IT department.

The implementation of the intraoperative frontal EEG monitoring performed routinely in this type of operation does not prolong the duration of the anesthesia. The placement and adjustments of the O3 or Foresight electrode and the transcranial Doppler probe takes only 5 to 10 minutes.

The physician in charge of the study collecting the data does not participate at any time in the management of the patient. The measures cannot influence the prescribing physician since at this stage the data are not yet analyzed and available.

The main objective is to identify a significant linear relationship between the percentage change in Vm and the percentage change in the 95% spectral frequency front (SEF95) during the MAP change.

The objective is to reject the null hypothesis based on the R2 measure of goodness of fit: H0: R2 = 0.

Considering a type I error probability = 0.05 and a power of 85%, and an effect size of 0.3 based on preliminary data. For a single predictor, the physician obtain a sample size of n = 32 patients. To adjust for possible confounding factors, the physician assume a partial correlation coefficient rho=0.5 between Vm and the covariates. This correction gives us a sample size of 32*2 = 64 patients (11). Finally, preliminary data indicate that 30% of the included patients have a poor signal or defective measurements resulting from artifacts or unsuitable experimental conditions. The final number of patients to be included is estimated at N = 100.

Rejection of the primary null hypothesis will be established by a linear regression model.

As a secondary objective, linear regression will also be evaluated between Vm and EEG markers such as alpha band power, time spent in burst-suppression, and delta-to-alpha ratio.

Descriptive statistics will be reported as n (%) for categorical variables, mean(standard deviation) for continuous variables, and median[IQR] for ordinal variables that do not have a normal distribution.

All statistical analyses will be performed using R statistical software (The 'R' Foundation for Statistical Computing, Vienna, Austria). Results will be expressed as means (± standard deviation). A p-value of less than 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age (≥ 18 years)
* Eligible for scheduled surgery at Lariboisière Hospital
* Informed patient who has expressed no objection to participating in this research

Exclusion Criteria:

* Patients under 18 years of age.
* Patient opposed to participation in the protocol
* Pregnant woman
* Patient under judicial protection
* Patient not affiliated to a social health system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery under general anesthesia with an intravenous anesthesia protocol with a concentration target (Orchestra® Base Primea - Fresenius Kabi France), a vasopressor support by norepinephrine and blood pressure optimisation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
mean arterial pressure | 1 day
  Continuous non-invasive measurement of mean arterial pressure (MAP, mmHg)
cerebral blood velocity in the middle cerebral artery | 1 day
  Measurement of cerebral blood velocity in the middle cerebral artery by Transcranial Pulsed Doppler. This corresponds to the Mean velocity (Vm) expressed in cm/s.
burst suppression | 1 day
  Continuous measurement of burst suppression (BS) (%)
95% spectral frequency front | 1 day
  Continuous measurement of a 95% spectral frequency front (SEF95) on the frontal EEG
delivered doses of hypnotics, morphine and paralytic agents | 1 day
  Quantification of delivered doses of hypnotics, morphine and paralytic agents

SECONDARY OUTCOMES:
Cerebral O2 saturation | 1 day
  Continuous measurement of cerebral O2 saturation (%) by near infraRed spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Fabrice VALLEE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Joaquim MATEO, Paris, France

IPD SHARING:
Plan to Share IPD: No